CLINICAL TRIAL: NCT05324709
Title: Yoga on Stress Management in Adolescents: Randomized Controlled Trial
Brief Title: Yoga on Stress Management in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, nesrin arslan, Principal Investigator, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-799
Record Dates: First submitted 2022-03-17; First posted 2022-04-12 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Adolescent Behavior; Adolescent Problem Behavior
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The program will be carried out one day a week for four weeks. Yin yoga practices will be applied in the program. Each session will last a total of 40 minutes. The first 20 minutes of yin yoga sessions. Participants will be given training on stress management, breathing and yin yoga. Afterwards, each session of Yin yoga exercises will be started with pranayama (breathing) exercises for 2 minutes, followed by Suryanamaskar-A (Sun Salute-A) for warming up and Yin yoga exercises will be done. The program will be completed by applying the focus on Moment in the last 5 minute. In addition, the participants will be given homework related to the subject of each week. The training booklet will be distributed to the participants before the program. Stress management sessions of the Adolescent Health Promotion-Physical Activity, Nutrition, Stress Management (COPE HEALTH- TEEN ) program will be used in the stress management training to be explained in the program.
  Interventions: Behavioral: Yoga Based Stress Management Program
- No Intervention (No Intervention): The control group will be given 60 minutes of "in the moment" and stress management training.

INTERVENTIONS:
Behavioral: Yoga Based Stress Management Program — Yoga-based stress management program is applied to the intervention group.
  Arms: Experimental

SUMMARY:
The World Health Organization (WHO, 2013) defined the 10-19 age group as "adolescent" and the 15-24 age group as "youth". Adolescence period; It is a period of rapid growth, development and maturation in terms of physical, mental, biochemical and social aspects.10-20% of children and adolescents living in the world have mental health diseases such as generalized anxiety disorders, depression, eating disorders, and post-traumatic stress disorders.In adolescents, yoga is practiced as a relaxing tool to reduce stress, especially for exam anxiety.In Turkey, there are no yoga-based experimental studies to prevent anxiety, stress and depression in adolescents.

DETAILED DESCRIPTION:
The aim of the study is to examine the effect of the Yoga-Based Stress Management Program on the ability to cope with stress in adolescents.Stress management sessions of the Adolescent Health Promotion-Physical Activity, Nutrition, Stress Management (COPE HEALTH-TEEN) program will be used in the stress management training to be explained in the program. There will also be yin yoga exercises.

The general population of the research will be high school senior students in Safranbolu district of Karabük province in the 2021-2022 academic year. First of all, the stress, anxiety and depression levels of the adolescents will be calculated. The research will be carried out in a total of 14 high schools. Each school will be determined as a "cluster" and 7 experimental and 7 control schools will be randomly selected. Simple random draw method will be applied in the selection of experimental and control schools. Adolescents who meet the inclusion criteria will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* High school senior student

  * Those who volunteered to participate in the research and
  * Students who are allowed to participate in the research by their parents

Exclusion Criteria:

* Students with any physical or mental disability • Low levels of perceived stress, anxiety, depression

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Change in stress level compared to baseline at 3 months. | Basaline, week 1, month 3
  Stress symptoms experienced by adolescents will be measured by the Perceived Stress Scale. A minimum of 0 and a maximum of 56 points are obtained from the scale. The high total score indicates the high level of stress experienced by the person.
Change in anxiety level compared to baseline at 3 months. | Basaline, week 1, month 3
  Anxiety symptoms experienced by adolescents will be measured with the Beck Anxiety Scale. A minimum score of 0 and a maximum of 63 points is obtained from the scale. The high total score indicates the high level of anxiety experienced by the person.
Change in depression level compared to baseline at 3 months. | Basaline, week 1, month 3
  Depression symptoms experienced by adolescents will be measured with the Reynolds Adolescent Depression Scale. A minimum of 30 and a maximum of 120 points can be obtained from the scale. A high total score indicates that the depression experienced by the person is high.

CONTACTS AND LOCATIONS:
Locations (1):
- Karabuk University, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No